CLINICAL TRIAL: NCT02358642
Title: A Randomized Placebo Controlled Trial of Low Dose Angiotensin Converting Enzyme Inhibitor to Prevent Pneumonia in Older People Who Require Tube Feeding Because of Neurological Dysphagia
Brief Title: Drug to Prevent Pneumonia in the Tube Fed
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The interim analysis suggested that low dose lisinopril given to be tube fed older patients with neuroligical dysphagia had increased mortality.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Department of Medicien and Therapeutics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACEI-RCT
Record Dates: First submitted 2013-02-28; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Pneumonia; Neurological Dysphagia
Keywords: Rate of Pneumonia; Mortality rate
MeSH Terms: conditions — Pneumonia | interventions — Angiotensin-Converting Enzyme Inhibitors; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Angiotensin converting enzyme inhibitor (Experimental): Angiotensin converting enzyme inhibitor (Lisinopril), 2.5mg, nocte, 26 weeks
  Interventions: Drug: Angiotensin converting enzyme inhibitor (Lisinopril)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Angiotensin converting enzyme inhibitor (Lisinopril)
  Arms: Angiotensin converting enzyme inhibitor
Drug: Placebo
  Arms: Placebo

SUMMARY:
Background: Older people with neurological dysphagia are at risk of recurrent aspiration pneumonia. Angiotensin converting enzyme inhibitor (ACEI) has been shown to improve swallowing and cough reflexes which may protect dysphagic patients from aspiration pneumonia.

Hypotheses: ACEI reduces the risk of pneumonia in older patients who are nasogastric tube fed because of dysphagia from cerebrovascular diseases.

Design: Randomized placebo controlled trial

Method: 302 older patients who have been tube fed for more than two weeks because of dysphagia secondary to cerebrovascular diseases are randomized to take half of lisinopril 5 mg or placebo tablet once daily for 26 weeks. The subjects will be recruited from medical wards in Prince of Wales and Shatin Hospitals, and from outpatients of geriatric or speech therapy clinics, who have had hospital stay in previous three months. The subjects are followed up at week 12 and 26. The primary outcome is the incidence rate of pneumonia as determined by pneumonic change on X ray and clinical criteria. The secondary outcomes are mortality rate, total episodes of pneumonia over 26 weeks, and swallowing ability defined by the Royal Brisbane Hospital Outcome Measure at week 12. Cost effectiveness analysis of public health care and personal health care costs will be performed. Intention to treat and log rank will be used to analyzed the group differences in outcomes. 60 subjects (30 in each trial group) recruited from medical inpatients at Prince of Wales Hospital will undergo swallowing videofluoscopy at baseline and week 12 follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Tube fed for more than four weeks for reason of neurological dysphagia as recommended by a trained speech therapist;
* clinical diagnosis of cerebrovascular diseases, confirmed by CT head scan. The reason for restricting the subjects to those with cerebrovascular disease is that previous studies which showed beneficial effects of ACEI on dysphagia were mostly based on stroke patients.

Exclusion Criteria:

* life expectancy less than six months;
* live outside Shatin area;
* systolic blood pressure less than 100 mm Hg;
* known intolerance of ACEI;
* existing use of ACEI or angiotensin receptor blockers;
* symptomatic chronic lung disease or cardiac failure;
* frequent withdrawal of enteral tube by patients;
* serum creatinine >100 µmol/L;
* serum potassium > 5.1 mmol/L.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence rate of pneumonia | week 26

SECONDARY OUTCOMES:
Number of pneumonia episodes | week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong